CLINICAL TRIAL: NCT04994652
Title: A Randomised Trial of Videolaryngoscopy Or Direct Laryngoscopy for Endotracheal Intubation in Newborn Infants
Brief Title: Video- Or Direct Laryngoscopy for Endotracheal Intubation in Newborns
Acronym: VODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VODE01
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Intubation, Intratracheal; Infant, Newborn; Laryngoscopes

STUDY DESIGN:
Intervention Model Description: Parallel group, randomised clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videolaryngoscope (Experimental): Intubation attempted with C-MAC videolaryngoscope
  Interventions: Device: Videolaryngoscopy
- Standard laryngoscope (Active Comparator): Intubation attempted with standard laryngoscope
  Interventions: Device: Direct laryngoscopy

INTERVENTIONS:
Device: Videolaryngoscopy — Indirect laryngoscopy using the C-MAC videolaryngoscope
  Arms: Videolaryngoscope
Device: Direct laryngoscopy — Direct laryngoscopy with a standard laryngoscope
  Arms: Standard laryngoscope

SUMMARY:
Endotracheal intubation is a critical intervention for newborn babies. Laryngoscopy is the crucial part of endotracheal intubation. Traditionally, operators use a standard laryngoscope to view the larynx by looking directly into the mouth (direct laryngoscopy). More recently videolaryngoscopes that have a video camera mounted at the tip of the laryngoscope blade have been developed, Rather than look directly into the mouth, the operator looks at a screen that displays the view acquired by the camera (indirect laryngoscopy). Videolaryngoscopes have been demonstrated to be useful for teaching trainees direct laryngoscopy. However, it may be that all clinicians are more successful with a videolaryngoscope. The investigators will compare whether clinicians who are randomly assigned to intubate newborn infants using a videolaryngoscope are more successful in intubating newborn infants at the first attempt compared to clinicians who are randomly assigned to intubate newborn infants using a standard laryngoscope.

DETAILED DESCRIPTION:
Endotracheal intubation is a critical intervention for newborn babies. Proficiency at intubation has declined markedly in recent decades such that fewer than half of babies are successfully intubated at the first attempt. Laryngoscopy is the crucial part of endotracheal intubation. Traditionally, operators use a standard laryngoscope to view the larynx by looking directly into the mouth (direct laryngoscopy). More recently videolaryngoscopes that have a video camera mounted at the tip of the laryngoscope blade have been developed, Rather than look directly into the mouth, the operator looks at a screen that displays the view acquired by the camera (indirect laryngoscopy). Videolaryngoscopes have been demonstrated to be useful for teaching trainees direct laryngoscopy, i.e. a senior colleague can coach them during the procedure. However, it may be that all clinicians are more successful with a videolaryngoscope. We will compare whether clinicians who are randomly assigned to intubate newborn infants using a videolaryngoscope are more successful in intubating newborn infants at the first attempt compared to clinicians who are randomly assigned to intubate newborn infants using a standard laryngoscope.

The investigators will study newborn infants who are undergoing intubation at the discretion of their treating clinicians in delivery room or in the Neonatal Intensive Care Unit (NICU).Term and preterm infants of any gender will be eligible to participate. Babies with upper airway anomalies will be ineligible. Participants will be randomly assigned in a 1:1 ratio to "VIDEO" or ""STANDARD" group. Intubation success will be determined in both groups using an exhaled carbon dioxide detector or flow sensor. Caregivers and outcome assessors will not be masked to group assignment. The investigators will enrol 214 babies to the study.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants (term and preterm, of any gender) in whom endotracheal intubation is attempted in the course of their clinical care in the Delivery Room or Neonatal Intensive Care Unit.

Exclusion Criteria:

* Infants with upper airway anomalies

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Intubation success at first attempt | 5 minutes
  Endotracheal intubation at first attempt confirmed with an exhaled carbon dioxide detector or flow sensor

SECONDARY OUTCOMES:
Lowest SpO2 during first intubation attempt | 5 minutes
  Lowest oxygen saturation recorded during first intubation attempt
Lowest HR during first intubation attempt | 5 minutes
  Lowest heart rate during first intubation during first intubation attempt
Number of attempts taken to intubate successfully | 30 minutes
  Number of attempts taken to successfully intubate the infant
Duration of successful attempt | 30 minutes
  Interval measured in seconds from the introduction of the laryngosocpe blade into the infants mouth to its removal in the successful intubation attempt
Crossover to alternative device | 30 minutes
  Use of alternative non-assigned laryngosocpe to attempt intubation
Correct ETT tip position on CXR | 1 hour
  Correct endotracheal tube tip position (i.e. between upper border of first thoracic vertebra and lower border of second thoracic vertebra) on chest radiograph

CONTACTS AND LOCATIONS:
Locations (1):
- National Maternity Hospital, Dublin, Co. Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Reasonable requests to share IPD will be considered
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Geraghty LE, Dunne EA, Ni Chathasaigh CM, Vellinga A, Adams NC, O'Currain EM, McCarthy LK, O'Donnell CPF. Video versus Direct Laryngoscopy for Urgent Intubation of Newborn Infants. N Engl J Med. 2024 May 30;390(20):1885-1894. doi: 10.1056/NEJMoa2402785. Epub 2024 May 5. PMID 38709215